CLINICAL TRIAL: NCT05240508
Title: Platelet FcGammaRIIa and Risk of Venous Thromboembolism in Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Chris Holmes, Professor of Medicine, University of Vermont
Other Study IDs: 1R21CA267074 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Venous Thromboembolism
Keywords: Platelet; Cancer
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thrombosis is common and contributes significantly to morbidity and mortality in patients with cancer. At least 20% of patients with cancer develop venous thromboembolism (VTE) and another 5% will experience acute arterial thromboembolism (ATE) due to cancer and its treatment. Current guidelines recommend VTE thromboprophylaxis in high-risk outpatients. Thromboprophylaxis strategies are inadequate as 50% of high-risk patients on prophylaxis still develop a VTE, the rate of recurrent VTE is ~24% with a case fatality rate of 14.8%, and the incidence of major bleeding is ~13% with a case fatality rate of 8.9%. We and others have implicated platelets in both the pathogenesis of VTE as well as cancer growth and metastasis. To investigate a new biomarker of risk in patients with cancer, we propose a pilot study to determine whether quantification of platelet FcɣRIIa expression can discriminate risk of VTE and cancer progression. We chose platelet FcɣRIIa expression because we have found that quantifying platelet surface expression of FcγRIIa identifies patients at high and low risk of thrombotic arterial events. Thus, we hypothesize that elevated platelet expression of FcγRIIa will identify patients with cancer who are greater risk of VTE as well as cancer progression. The proposed studies leverage a clinical research program that was established in 2015 at the University of Vermont Cancer Center (Venous Thromboembolism Prevention in the Ambulatory Care Clinic [VTEPACC]) and will allow simultaneous access to research samples, thrombosis complications and cancer outcomes in order to achieve the following specific aims: 1) To determine whether platelet expression of FcγRIIa identifies cancer patients at high and low risk of VTE, and 2) To determine whether increased platelet expression of FcγRIIa is associated with a) advanced stage cancer at the time of enrollment and b) greater progression of cancer. Platelet reactivity is increased in patients with cancer and has been associated with VTE risk. Platelet expression of FcγRIIa can increase the risk of thrombosis by both increasing platelet reactivity and by promoting the procoagulant potential of platelets. In addition, platelets promote cancer by facilitating tumor vascularization, growth, and metastasis. FcγRIIa has been shown to be a key mediator of platelet secretion and cross-talk between platelets and tumor cells. Thus, we propose that increased platelet FcγRIIa expression will be linked to enhanced tumor growth and metastasis by facilitating cancer-tumor cell cross-talk and thereby the activation of platelets that leads to the release of platelet products. Identification of a biomarker capable of discriminating high and low risk of VTE will provide an important precision tool that could be combined with existing tools to guide therapy and improve outcomes. Results from aim 2 will provide key preliminary data in support of novel antiplatelet treatments to limit cancer progression.

ELIGIBILITY:
Inclusion Criteria:

* Active cancer diagnosis receiving cancer directed therapy
* Willing to consent to participation

Exclusion Criteria:

* unwilling to provide informed consent,
* clinical or study physician declines patient enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a cancer diagnosis who are anticipating starting new outpatient directed chemotherapy/immunotherapy/hormonal or biologic therapy or who will be changing therapy due to disease progression or relapse.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
venous thromboembolism occurrence | 18 months
  development of VTE or PE
Cancer Progression | 18 months
  Progression and stage of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Chris Holmes, MD PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States